CLINICAL TRIAL: NCT02389309
Title: A Phase I Trial of Dasatinib (PDGFR and SRC Inhibitor), Temsirolimus, and Cyclophosphamide in Patients With Advanced Solid Tumors
Brief Title: Dasatinib, Temsirolimus, and Cyclophosphamide in Treating Patients With Advanced, Recurrent, or Refractory Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0692; NCI-2015-00524 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-0692 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2015-03-04; First posted 2015-03-17 (Estimated); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Advanced Malignant Solid Neoplasm; Recurrent Brain Neoplasm; Recurrent Malignant Solid Neoplasm; Refractory Brain Neoplasm
MeSH Terms: conditions — Brain Neoplasms | interventions — Cyclophosphamide; Dasatinib; temsirolimus; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (dasatinib, cyclophosphamide, temsirolimus) (Experimental): Patients receive dasatinib PO BID on days 1-21, cyclophosphamide PO QD on days 1-21, and temsirolimus IV over 30-60 minutes on days 1, 8, and 15. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients experiencing stable disease or better may continue treatment with the approval of the Study Chair.
  Interventions: Drug: Cyclophosphamide; Drug: Dasatinib; Other: Laboratory Biomarker Analysis; Drug: Temsirolimus

INTERVENTIONS:
Drug: Cyclophosphamide — Given PO
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Dasatinib — Given PO
  Other Names: BMS-354825; Sprycel
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Temsirolimus — Given IV
  Other Names: CCI-779; CCI-779 Rapamycin Analog; Cell Cycle Inhibitor 779; Rapamycin Analog; Rapamycin Analog CCI-779; Torisel

SUMMARY:
This phase I trial studies the side effects and best dose of dasatinib and temsirolimus when given together with cyclophosphamide in treating patients with solid tumors that have spread to other places in the body, have come back, or have not respond to previous treatment. Dasatinib and temsirolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as cyclophosphamide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving dasatinib and temsirolimus together with cyclophosphamide may be a better treatment for advanced solid tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) and dose-limiting toxicities (DLT) of combination treatment with dasatinib, cyclophosphamide and temsirolimus.

II. To define and describe the toxicities of the combination of dasatinib, cyclophosphamide and temsirolimus administered on this schedule.

SECONDARY OBJECTIVES:

I. To preliminarily define the antitumor activity of the combination of dasatinib, cyclophosphamide and temsirolimus within the confines of a phase 1 study.

II. Preliminary assessment of biological markers and correlates of response.

OUTLINE: This is a dose-escalation study of dasatinib and temsirolimus.

Patients receive dasatinib orally (PO) twice daily (BID) on days 1-21, cyclophosphamide PO once daily (QD) on days 1-21, and temsirolimus intravenously (IV) over 30-60 minutes on days 1, 8, and 15. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients experiencing stable disease or better may continue treatment with the approval of the study chair.

After completion of study treatment, patients are followed up for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be >/= 12 months and < 21 years of age at the time of study enrollment.
* Patients must have had a previous histological verification of a solid tumor at the original diagnosis and/or recurrence including brain tumors; for patients with brain stem gliomas and optic pathway tumors, the requirement for histological evaluation may be waived; the patient's disease must be considered refractory to conventional/standard therapy, or a disease for which no conventional therapy exists and is progressive
* The patient must have a stable clinical (neurologic in case of brain tumors) exam and be on a stable dose of steroids for at least 1 week prior to study entry; the patient should have a measurable and/or evaluable disease; measurable disease which is defined as the presence of at least one lesion that can be accurately measured in two dimensions (each measures at least 10 mm) or evaluable disease which is defined as at least one lesion that can be accurately measured in at least one dimension (measure at least 10 mm)
* Karnofsky performance status >= 50 for patients >= 16 years of age and a Lansky performance status >= 50 for patients aged < 16 years
* Life expectancy: must be >= 12 weeks
* Chemotherapy:

  * Must not have received myelosuppressive chemotherapy within 3 weeks of the study entry (6 weeks if prior nitrosourea); prior treatment with either dasatinib or temsirolimus but not both is allowed; at least 3 weeks must have elapsed from the last dose
* Biologic therapy (anti-neoplastic)

  * Must not have received oral tyrosine kinase inhibitors (other than dasatinib) or other similar agents within 3 weeks of the study entry and all toxicities must have resolved to < grade 2 prior to enrollment
  * Must not have received bevacizumab or other monoclonal antibody therapy within 4 weeks of study the entry
* Radiotherapy (XRT): at least 4 weeks for focal XRT or 8 weeks for craniospinal XRT must have elapsed prior to study entry
* Stem cell transplant (SCT): at least 8 weeks following autologous SCT and 12 weeks for allogeneic SCT
* Surgery: at least 2 weeks following surgery including brain and spine provided post-operative magnetic resonance imaging (MRI) shows no active bleeding
* Concomitant medications: the following drugs need to be stopped at the time of beginning therapy: patient cannot be on liver enzyme inducing anticonvulsants; patients must not have received growth factors to support the number or function of white cells or platelets within the past 7 days and pegfilgrastim within the past 14 days; patients must not be receiving any anti-thrombotic or anti-platelet agents; patient cannot be on drugs that cause significant prolonged QT (category I drug)
* Absolute neutrophil count (ANC) greater than or equal to 1000/mm^3
* Platelets greater than or equal to 75,000/mm^3 (transfusion independent; no transfusion for >= 7 days prior to study enrollment)
* Hemoglobin greater than 8.0 g/dL (transfusion independent; no transfusion for >= 7 days prior to study enrollment)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 3 x upper limit of normal for age (ULN)
* Bilirubin =< 1.5 x ULN
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) > 70 ml/min/1.73 m^2 OR serum creatinine based on age/gender as follows:

  * Age 1 to < 2 years, 0.6 mg/dL (male) and 0.6 mg/dL (female)
  * Age > 2 and < 6 years, 0.8 mg/dL(male) and 0.8 mg/dL (female)
  * Age > 6 and < 10 years, 1.0 mg/dL (male) and 1.0 mg/dL (female)
  * Age > 10 and < 13 years, 1.2 mg/dL (male) and 1.2 mg/dL (female)
  * Age > 13 and < 16 years, 1.5 mg/dL (male) and 1.4 mg/dL (female)
  * Age > 16 years, 1.7 mg/dL (male) and 1.4 mg/dL (female)
* All post-menarchal females must have a negative serum beta-human chorionic gonadotropin (beta HCG); sexually active patients of childbearing potential must agree to use an effective method of contraception during the study and for at least 6 months after
* Adequate pulmonary function as defined as: no evidence of dyspnea at rest, no exercise intolerance, and a pulse oximetry > 94% if there is clinical indication for determination
* Adequate cardiac function defined as: normal 12 lead electrocardiogram (EKG) with corrected QT interval (QTc) < 450 msec, and either shortening fraction of >= 28% by echocardiogram and qualitatively normal left ventricular function, or ejection fraction of >= 55% by echocardiogram
* Patients with seizure disorder may be enrolled if on non-enzyme inducing anticonvulsants and well controlled
* Serum cholesterol and serum triglyceride levels must be < grade 2
* A written informed consent MUST be obtained from the patients and/or their parents/legal guardians prior to enrollment indicating their awareness of investigational nature of this study

Exclusion Criteria:

* Patients with evidence of recent intratumoral hemorrhage (within 3 months of study enrollment), gastrointestinal bleeding, history of coronary artery disease or on anticoagulation therapy
* Pregnant or breast-feeding women will not be entered on this study
* Uncontrolled current illness including, but not limited to, uncontrolled infection, need for hemodialysis, need for ventilatory support, psychiatric illness/social situations that would limit compliance with study requirements
* History of hypersensitivity to any component of the formulation
* Patients with known human immunodeficiency virus (HIV) are ineligible for this study
* Patients must not have received prior therapy with dasatinib and temsirolimus for any indication
* Patients with clinically significant cardiovascular disease: history of ischemic or hemorrhagic stroke within past 6 months; uncontrolled hypertension, on at least 2 repeated determinations on separate days within past 3 months; myocardial infarction or unstable angina within past 6 months; New York Heart Association grade III or greater congestive heart failure, serious cardiac arrhythmia requiring medication, unstable angina pectoris within past 6 months; clinically significant peripheral vascular disease within past 6 months; pulmonary embolism, deep vein thrombosis (DVT), or other thromboembolic event within past 6 months; diagnosed congenital long QT syndrome; any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or torsades de pointes); prolonged QTc interval on pre-entry electrocardiogram (> 450 msec); subjects with hypokalemia or hypomagnesemia if it cannot be corrected prior to dasatinib administration
* Anticonvulsants: patients on enzyme inducing anticonvulsants (EIAED) will be excluded; if patients were previously on EIAEDs that have been discontinued, patients must have been off EIAEDs for >= 2 weeks prior to initiation of dasatinib
* Anticoagulants/anti-platelets: patients on therapeutic (treatment) dose of anticoagulants (e.g. warfarin, low molecular-weight heparin) are not eligible; patients are not allowed to take aspirin, clopidogrel, ticlopidine, Aggrenox; patients on prophylactic anticoagulation may be enrolled and treated on study as long as their platelet count is monitored closely and maintained at > 75,000 while they are receiving dasatinib
* Inducers and Inhibitors of cytochrome P450 family 3, subfamily A, polypeptide 4 (CYP3A4): patients required to be on any CYP3A4/5 inhibitors or inducers will be excluded (with the exception of dexamethasone, but all efforts should be made to reduce the dose of dexamethasone); patients must discontinue drug at least 7 days prior to starting dasatinib
* Angiotensin-converting enzyme (ACE) inhibitors: patients who are currently receiving ACE inhibitors are not eligible
* Anti-graft-versus-host disease (GVHD) or agents to prevent organ rejection post-transplant: patients who are receiving cyclosporine, tacrolimus or other agents to prevent either graft-versus-host disease post bone marrow transplant or organ rejection post-transplant are not eligible for this trial
* Category I drugs that are generally accepted to have a risk of causing torsades de pointes including: (patients must discontinue drug at least 7 days prior to starting dasatinib)

  * Quinidine, procainamide, disopyramide
  * Amiodarone, sotalol, ibutilide, dofetilide
  * Chlorpromazine, haloperidol, mesoridazine, thioridazine, pimozide
  * Cisapride, bepridil, droperidol, arsenic, chloroquine, domperidone, halofantrine, levomethadyl, sparfloxacin, lidoflazine
* Other drugs permitted but use with caution include; drugs are not recommended but can be used with caution

  * Antacids: use of H2 blockers and proton pump inhibitors is not recommended; patients who require antacids should use short acting, locally active agents (e.g., Maalox, Mylanta etc.); however, these agents should not be taken within either 2 hours before or 2 hours after the dasatinib dose
  * Drugs prolong QT interval; erythromycin, clarithromycin, pentamidine, ondansetron, granisetron, and methadone

Ages: 12 Months to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2015-10-05 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) defined as the highest dose level tested at which =< 2/6 patients experience dose limiting toxicities (DLT) graded according to the National Cancer Institute (NCI) Common Toxicity Criteria (CTCAE) version 4.0 | Up to day 35
Incidence of adverse events (AEs) graded according to NCI CTCAE version 4.0 | Up to 28 days post-treatment
  AEs will be tabulated by dose, grade, and attribution.

SECONDARY OUTCOMES:
Best response (complete response [CR], partial response [PR], stable disease [SD], and progressive disease [PD]) using the Response Evaluation Criteria in Solid Tumors from the NCI for assessment of radiographic response | Up to 4 weeks post-treatment
  Tabulated by dose and disease category (CR, PR, SD, and PD).
Levels of biological markers measured in tissue, blood, or plasma | Up to 4 weeks post-treatment
  Correlation of biomarkers between tissue and blood will be assessed. The association among various continuous and discrete variables (including response variable) will be assessed first by the exploratory data analysis graphically and then tested using t-test/analysis of variance or Wilcoxon rank sum test/Kruskal-Wallis test, when appropriate. Correlation among continuous biomarkers will be examined by Pearson or Spearman rank correlation coefficients. The association between discrete variables will be tested by chi-square or Fisher's exact test.

CONTACTS AND LOCATIONS:
Overall Officials: Wafik T Zaky, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org